CLINICAL TRIAL: NCT07237711
Title: Clinical Investigation of Sensovisc Sterile Sodium Hyaluronate Gel in the Knee Joint
Brief Title: Clinical Investigation of Sensovisc
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Collaborators: İstem Medikal Tıbbi Cihaz ve Sanayi Ticaret Anonim Şirketi (Unknown)
Responsible Party: Principal Investigator, Emre Adıgüzel, Prof. MD, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AnkaraCHBilkentHayriyesimsek02
Record Dates: First submitted 2025-11-14; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Osteo Arthritis of the Knee
Keywords: viscosupplementation; knee osteoarthritis; hyaluronic acid; dosing; Sensovisc
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Injections, Intra-Articular

STUDY DESIGN:
Intervention Model Description: Patients are randomised to receive varying dosing regimens of Sensovisc
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SV-2-40 or SV-3-60 (Experimental): Patients with a Visual Analogue Scale (VAS) score of 80 mm or higher will receive a single injection of SV-3-60 (Sterile Sodium Hyaluronate Gel-3 mL Prefilled Syringe (2.0%)), whereas those with a score below 80 mm will receive a single injection of SV-2-40 (Sterile Sodium Hyaluronate Gel-2 mL Prefilled Syringe (2.0%) )
  Interventions: Device: Sensovisc®
- SV-2-32 (Experimental): For the patients who will be injected with SV-2-32 (Sterile Sodium Hyaluronate Gel-2 mL Prefilled Syringe (1.6%)), a second injection will be performed 1 week after the first injection.
  Interventions: Device: Sensovisc®
- SV-2-20 (Experimental): 3 intra-articular injections of SV-2-20 (Sterile Sodium Hyaluronate Gel-2 mL Prefilled Syringe (1.0%)) administered 1 weeks apart. For the subject in the SV-2-20 group, a second and third injection will be performed one week and two weeks after the first injection.
  Interventions: Device: Sensovisc®

INTERVENTIONS:
Device: Sensovisc® — Injectable Sterile Sodium Hyaluronate Gel
  Other Names: Hyaluronic Acid Gel; Intra-articular injection; Sodium Hyaluronate

SUMMARY:
This clinical investigation aims to investigate the safety and performance of Sensovisc.

Sensovisc is used to reduce osteoarthritis (OA) related pain in the joints by supporting synovial fluid by intra-articular injection and allowing the synovial fluid to restore its viscoelastic properties. It increases the joint mobility by reducing or eliminating the pain.

This Clinical Investigation was designed as a cross-sectional, interventional, and prospective study.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most prevalent chronic arthritis and a leading cause of pain and disability among adults. OA is a degenerative joint disease characterized by chronic inflammation, cartilage degradation and erosion of underlying bone in the affected joints, predominantly affects knees, significantly impacting patient mobility and quality of life.

* Although there are currently no approved disease-modifying osteoarthritis drugs (DMOADs), nonpharmacologic interventions, such as physical therapy and weight management, and pharmaceutical approaches are available to reduce or revise joint damage and inflammation.
* Among various therapeutic interventions, intra-articular hyaluronic acid (HA) injections have emerged as an alternative promising treatment. Emerging evidence suggests that HA may exert chondroprotective effects by enhancing synovial fluid viscosity, improving joint lubrication, and mitigating inflammatory processes, thereby potentially decelerating disease progression and preserving cartilage integrity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have unilateral and/or bilateral knee pain for more than 3 months and meet the diagnosis of osteoarthritis according to ACR criteria
* Diagnosis of Stage II or III knee OA according to the Kellgren and Lawrence (K&L) classification, determined by x-rays taken in the last 12 months
* 40 mm above the pain level determined by VAS during rest for at least 15 days in the month before starting the study (for paracetamol and oral nonsteroidal anti-inflammatory drugs (NSAIDs), taking into account the half-life of the drug)
* Having a Body Mass Index (BMI) ≤ 40 kg/m²,
* Having the mental ability to express pain scores
* Signing the informed consent form indicating consent to participate in the study

Exclusion Criteria:

* Radiological K&L stage I and IV
* Acute inflammatory osteoarthritis attack (KOFUS ≥7)
* Septic arthritis
* Secondary OA [Synovial chondromatosis or pigmented villonodular synovitis of the knee, Joint diseases (joint dysplasia, aseptic osteonecrosis, acromegaly, Paget's disease, hemophilia, hemochromatosis), Inflammatory diseases (rheumatoid arthritis, gout, infectious arthritis, acute calcium pyrophosphate arthritis)]
* Ipsilateral cruciate or collateral ligament injury in the last 3 months,
* Corticosteroid injection into the target knee within the last 1 month before the first injection
* Hyaluronat injection into the target knee within the last 6 months before the first injection
* Arthroscopy or surgery on the target knee within the last 6 months before the first injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2026-08-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Baseline
  VAS at rest: Measures pain intensity while resting. Scale 0-10 cm (0 = no pain, 10 = worst imaginable pain). Higher scores = worse pain at rest.
  VAS at night: Measures pain intensity during the night, especially disturbing sleep. Scale 0-10 cm. Higher scores = worse nocturnal pain.
  VAS during activity: Measures pain intensity during movement or activity. Scale 0-10 cm. Higher scores = worse pain on activity.
WOMAC Osteoarthritis Index | Baseline
  The WOMAC Index is a self-administered questionnaire designed to evaluate symptoms and functional limitations in hip and knee osteoarthritis. It has 3 subscales:
  Pain (0-20) Stiffness (0-8) Physical function (0-68) The total score ranges from 0 to 96, with higher scores indicating worse pain, stiffness, and functional impairment.
Lequesne's Algofunctional Index for Knee | Baseline
  It measures three areas:
  Pain/discomfort (during activities and at rest), Maximum walking distance Daily living activities (like standing up, climbing stairs, squatting) The total score ranges from 0 to 24, with higher scores indicating greater disability: 1-4 = mild, 5-7 = moderate, 8-10 = severe, ≥14 = extremely severe.
Change in Visual Analogue Scale (VAS) score from baseline at 6 weeks | 6 weeks after last injection
  VAS at rest: Measures pain intensity while resting. Scale 0-10 cm (0 = no pain, 10 = worst imaginable pain). Higher scores = worse pain at rest.
  VAS at night: Measures pain intensity during the night, especially disturbing sleep. Scale 0-10 cm. Higher scores = worse nocturnal pain.
  VAS during activity: Measures pain intensity during movement or activity. Scale 0-10 cm. Higher scores = worse pain on activity.
Change in WOMAC Osteoarthritis Score from baseline at 6 weeks | 6 weeks after last injection
  The WOMAC Index is a self-administered questionnaire designed to evaluate symptoms and functional limitations in hip and knee osteoarthritis. It has 3 subscales:
  Pain (0-20) Stiffness (0-8) Physical function (0-68) The total score ranges from 0 to 96, with higher scores indicating worse pain, stiffness, and functional impairment.
Change in Lequesne's Algofunctional Score from baseline at 6 weeks | 6 weeks after last injection
  It measures three areas:
  Pain/discomfort (during activities and at rest), Maximum walking distance Daily living activities (like standing up, climbing stairs, squatting) The total score ranges from 0 to 24, with higher scores indicating greater disability: 1-4 = mild, 5-7 = moderate, 8-10 = severe, ≥14 = extremely severe.
Change in Visual Analogue Scale (VAS) score from baseline at 6 months | 6 months after last injection
  VAS at rest: Measures pain intensity while resting. Scale 0-10 cm (0 = no pain, 10 = worst imaginable pain). Higher scores = worse pain at rest.
  VAS at night: Measures pain intensity during the night, especially disturbing sleep. Scale 0-10 cm. Higher scores = worse nocturnal pain.
  VAS during activity: Measures pain intensity during movement or activity. Scale 0-10 cm. Higher scores = worse pain on activity.
Change in WOMAC Osteoarthritis Score from baseline at 6 months | 6 months after last injection
  The WOMAC Index is a self-administered questionnaire designed to evaluate symptoms and functional limitations in hip and knee osteoarthritis. It has 3 subscales:
  Pain (0-20) Stiffness (0-8) Physical function (0-68) The total score ranges from 0 to 96, with higher scores indicating worse pain, stiffness, and functional impairment.
Change in Lequesne's Algofunctional Score from baseline at 6 months | 6 months after last injection
  It measures three areas:
  Pain/discomfort (during activities and at rest), Maximum walking distance Daily living activities (like standing up, climbing stairs, squatting) The total score ranges from 0 to 24, with higher scores indicating greater disability: 1-4 = mild, 5-7 = moderate, 8-10 = severe, ≥14 = extremely severe.

SECONDARY OUTCOMES:
The usability of the devices | Baseline
  Device usability will be evaluated using a structured, multidimensional Device Usability Assessment Form, which includes five domains:
  Evaluation of the Product Instructions for Use Evaluation of the Surgical Technique Guide Evaluation of the Implant Card Evaluation of the Operation (Syringe Handling and Injection Procedure) Evaluation of Packaging
  The assessment form contains Likert-type items rated on a 5-point scale:
  1 = Strongly disagree, 2 = Disagree, 3 = Neither agree nor disagree, 4 = Agree, 5 = Strongly agree.
  A higher score reflects better usability, easier handling, clearer instructions, and improved user satisfaction.